CLINICAL TRIAL: NCT01030016
Title: Blood Pressure Response During Resistance Exercise in Hypertensives: Influence of Beta-blockers
Brief Title: Study of Atenolol Influence on Blood Pressure During Resistance Exercise
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Cláudia Lúcia de Moraes Forjaz, School of Physical Education and Sport, University of São Paulo
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: FAPESP-06/06356-8
Record Dates: First submitted 2009-12-08; First posted 2009-12-10 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-05

CONDITIONS: Blood Pressure; Exercise
Keywords: resistance exercise; beta-blockers; blood pressure
MeSH Terms: conditions — Motor Activity | interventions — Atenolol; Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- atenolol (Experimental): subjects received 6 weeks of atenolol
  Interventions: Drug: atenolol

INTERVENTIONS:
Drug: atenolol — 25 mg/day, twice a day for 6 weeks
  Other Names: beta-blockers

SUMMARY:
The study was designed to investigate if atenolol is able to blunt blood pressure increase during resistance exercise in hypertensive subjects.

DETAILED DESCRIPTION:
The study compared intra-arterial blood pressure responses during leg-extension resistance exercise performed to fatigue at 40, 80 and 100% of 1 RM in hypertensive patients receiving placebo (first) and atenolol (second) on a single blind manner.

ELIGIBILITY:
Inclusion Criteria:

* hypertension with blood pressure levels below 160/105 mmHg under placebo.
* age between 30 and 60 years
* nonobese

Exclusion Criteria:

* target organ lesion
* cardiovascular risk factor
* cardiovascular disease
* physically active

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
blood pressure during resistance exercise | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cláudia LM Forjaz, PhD, Principal Investigator — University of Sao Paulo; Decio Mion Jr, PhD, Study Chair — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil